CLINICAL TRIAL: NCT02371772
Title: Comparison Between Conventional Anticoagulation Treatment and Self-management of Anticoagulation Treatment
Brief Title: Self-management of Anticoagulation Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Una Ørvim Sølvik (Other)
Responsible Party: Sponsor-Investigator, Una Ørvim Sølvik, Associate professor, University of Bergen
Organization: University of Bergen (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: UBergen
Record Dates: First submitted 2015-02-11; First posted 2015-02-26 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Long-term Oral Anticoagulant Therapy
Keywords: Warfarin; Self Care; Conventional care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-management anticoagulation treatment (Other): Trained to monitor INR and dose warfarin
  Interventions: Other: Training
- Conventional anticoagulation treatment (No Intervention): Before enrolment

INTERVENTIONS:
Other: Training — Patients were trained to monitor INR and dose warfarin
  Arms: Self-management anticoagulation treatment

SUMMARY:
The aim of the study was to compare self-management of anticoagulant treatment with conventional anticoagulant treatment in Norway.

DETAILED DESCRIPTION:
Patients (n=23) on anticoagulant treatment with warfarin participated in a 27 weeks training program where they learned how to analyse International Normalised Ratio (INR) using the point-of-care instrument CoaguChek® XS and dose warfarin. The patients had to display their skills through a test before considered self-managing. They continued to measure INR weekly for 28 weeks. All INR values during the training program and self-control period were collected. In addition, the patients were told to notify if they had any complications during this period. Ten INR values and complications before enrolment was collected from INR cards and/or their general practioner. The participant filled in a quality of life-questioner at enrolment and after 28 weeks of self-management.

ELIGIBILITY:
Inclusion Criteria:

* on life-long oral anticoagulation therapy
* Live in Bergen municipality
* Judged to be qualified for patient self-management anticoagulation treatment by their GP
* Motivated to follow the training program

Exclusion Criteria:

* Drug abuse
* Liver disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Change in Time in therapeutic range (TTR) | From 39 weeks before enrolment until 28 weeks of self management

SECONDARY OUTCOMES:
Change in number of complications | From 39 weeks before enrolment until 28 weeks of self management

CONTACTS AND LOCATIONS:
Overall Officials: Una Ø Sølvik, PhD, Principal Investigator — University of Bergen